CLINICAL TRIAL: NCT06168045
Title: Arterial Blood Pressure and Cerebral Tissue Oxygenation During Immediate Transition After Birth in Term and Preterm Neonates - a Prospective Pilot Observational Study
Brief Title: Bloodpressure and NIRS During the Immediate Transition
Acronym: RR
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Pichler Gerhard, MD., Prof, Medical University of Graz
Other Study IDs: 1026/2022 (34-221 ex 21/22)
Record Dates: First submitted 2023-11-23; First posted 2023-12-13 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Blood Pressure; Cerebral Tissue Oxygenation
MeSH Terms: interventions — Blood Pressure Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Term neonates: Neonates with gestational age 37+0 - 42+0 weeks
  Interventions: Diagnostic Test: Cerebral tissue oxygenation and blood pressure measurement
- Preterm neonates: Neonates with gestational age < 37+0 weeks
  Interventions: Diagnostic Test: Cerebral tissue oxygenation and blood pressure measurement

INTERVENTIONS:
Diagnostic Test: Cerebral tissue oxygenation and blood pressure measurement — Measurement of cerebral tissue oxygenation with NIRS and blood pressure during immediate transition after birth

SUMMARY:
Blood pressure will be measured in min. 5/10/15 after birth. Cerebral tissue oxygenation (crSO2) monitoring with NIRS in addition to routine arterial oxygen saturation (SpO2) monitoring with pulse oximetry will be performed continuously during the first 15 minutes after birth

ELIGIBILITY:
Inclusion Criteria:

Term and preterm neonates observed routinely immediately after birth at the resuscitation desk

* Decision to conduct full life support
* Written informed consent

Exclusion Criteria:

No decision to conduct full life support

* No written informed consent
* Congenital malformation

Ages: 1 Minute to 15 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Term and preterm neonates observed routinely at the resuscitation desk at the Division of Neonatology, Department of Pediatrics, Medical University of Graz will be eligible for the study.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 5, 10 and 15 minutes after birth
  Systolic, diastolic and mean blood pressure in mmHg measured with a pneumatic cuff
Cerebral oxygenation | 5, 10 and 15 minutes after birth
  Cerebral tissue oxygen saturation in percent measured with NIRS

SECONDARY OUTCOMES:
Cardiac output | 5, 10 and 15 minutes after birth
  Calculated out of blood pressure and heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Pichler, Prof, Principal Investigator — Medical University of Graz
Locations (1):
- medical university of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pichler G, Cheung PY, Aziz K, Urlesberger B, Schmolzer GM. How to monitor the brain during immediate neonatal transition and resuscitation? A systematic qualitative review of the literature. Neonatology. 2014;105(3):205-10. doi: 10.1159/000357162. Epub 2014 Jan 25. PMID 24481411
- [Background] Hooper SB, Te Pas AB, Lang J, van Vonderen JJ, Roehr CC, Kluckow M, Gill AW, Wallace EM, Polglase GR. Cardiovascular transition at birth: a physiological sequence. Pediatr Res. 2015 May;77(5):608-14. doi: 10.1038/pr.2015.21. Epub 2015 Feb 4. PMID 25671807
- [Background] Baik N, Urlesberger B, Schwaberger B, Avian A, Mileder L, Schmolzer GM, Pichler G. Blood Pressure during the Immediate Neonatal Transition: Is the Mean Arterial Blood Pressure Relevant for the Cerebral Regional Oxygenation? Neonatology. 2017;112(2):97-102. doi: 10.1159/000455965. Epub 2017 Apr 21. PMID 28427056

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT06168045/Prot_SAP_000.pdf